CLINICAL TRIAL: NCT07304128
Title: A Phase 1, Open-Label, Multi-Center, Dose Escalation and Expansion Study of PLB-002 (Anti-Claudin 6 ADC) in Adults With Advanced Solid Tumors
Brief Title: A Study of PLB-002 in Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Primelink BioTherapeitics(ShenZhen) Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PLB-002-001
Record Dates: First submitted 2025-12-01; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumor
Keywords: PLB-002; ovarian cancer; NSCLC; CLDN6; claudin6
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 2: Dose Expansion Study (Experimental): Patients with CLDN6 expression
  Interventions: Drug: PLB-002
- Part 1: Dose Escalation Study (Experimental): In the dose escalation part of the study, patients with advanced solid tumors will be treated with escalating doses of PLB-002.
  Interventions: Drug: PLB-002

INTERVENTIONS:
Drug: PLB-002 — antibody drug conjugate (ADC)

SUMMARY:
This study will test the safety, including side effects, and determine the characteristics of a drug called PLB-002 in participants with solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet all of the following criteria will be eligible to participate in the study:

  1. Patient must have the ability to understand and voluntarily sign a written informed consent form (ICF) and must have signed ICF prior to any study procedure.
  2. Adults aged 18 years or older.
  3. Histologically or cytologically confirmed advanced solid tumors, including platinum-resistant ovarian cancer (including fallopian tube and primary peritoneal carcinoma), NSCLC, testicular cancer, and other solid tumors, who have failed or intolerant to available standard-of-care therapy or no standard treatment exists.
  4. At least one measurable lesion as per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria.
  5. Performance status of Eastern Cooperative Oncology Group (ECOG) 0-1.
  6. Expected survival of 3 months or longer.
  7. Part 1: Available archived or fresh tissue for retrospective CLDN6 evaluation (patients in the backfill part are recommended to have positive CLDN6 staining results by immunohistochemistry [IHC] tested in the central laboratory before enrollment); Part 2: Positive CLDN6 staining of tumor tissue (archived or fresh) by IHC tested in the central laboratory.
  8. Have adequate organ function, as indicated by the following laboratory parameters in below table.

     Hematologic (no transfusion or hematopoietic stimulating factor treatment within 14 days) Neutrophils ≥ 1.5 × 109/L Platelets ≥ 100× 109/L Hemoglobin ≥ 90 g/L Hepatic function Total bilirubin ≤ 1.5×ULN (≤ 3.0×ULN for patients with Gilbert's syndrome or liver metastasis/ hepatocellular carcinoma) Alanine aminotransferase (ALT) ≤ 2.5×ULN (≤ 5.0×ULN for patients with liver metastasis/ hepatocellular carcinoma) Aspartate aminotransferase (AST) ≤ 2.5×ULN (≤ 5.0×ULN for patients with liver metastasis/ hepatocellular carcinoma) Albumin ≥ 3.0 g/dL Renal function Creatinine clearance (Ccr) ≥ 60 mL/min (Ccr calculated according to Cockcroft-Gault formula) Coagulation function Activated partial thromboplastin time (aPTT), international normalized ratio (INR) and prothrombin time ≤ 1.5 × ULN (If patients are receiving anticoagulant therapy: stable doses of anticoagulants must be taken for ≥ 1 month, and the prothrombin time/aPTT/INR must be within the intended therapeutic range) Cardiac function Left ventricular ejection fraction (LVEF) ≥ 50%
  9. Female patients should meet at least 1 of the following criteria before they can participate in the study:

     * Women of childbearing potential (WOCBP) must have a negative serum pregnancy test during the screening period (within 7 days prior to the first dose of the study drug), must not be lactating, and must be willing to practice a highly effective contraceptive method throughout the study (i.e., from study entry up to 6 months after the last dose of the study drug).
     * Females who have no childbearing potential (i.e., physiologically incapable of pregnancy), including those who have undergone hysterectomy, bilateral oophorectomy, or bilateral salpingectomy.
     * Postmenopausal (total cessation of menses for ≥ 1 year).
  10. Male patients are eligible to participate in the study if they have undergone a vasectomy or agree to use a highly effective method of contraception and refrain from donating sperm from study entry up to 6 months after the last dose of the study drug.

Exclusion Criteria:

* Patients who meet any of the following criteria will be excluded from participation in the study:

  1. Patient received systemic chemotherapy, small molecular target therapy, hormone therapy, or herbal medication with anti-cancer indication within 2 weeks prior to start of study drug; or received biological anti-cancer products (such as antibody, antibody-drug conjugate [ADC]) within 4 weeks or 5 half-life time prior to start of study drug (whichever is shorter). For cytotoxic agents with major delayed toxicity (such as nitrosourea or mitomycin C), 6 weeks of washout are mandated.
  2. Patients who have undergone radical radiotherapy within 4 weeks prior to the first dose of study drug, or have undergone brain stereotactic radiotherapy or whole brain radiotherapy within 4 weeks prior to the first dose of study drug, or have undergone palliative radiotherapy within 2 weeks prior to the first dose of study drug, or have used a radioactive drug (Strontium, Samarium, etc.) within 8 weeks prior to the first dose of the study drug.
  3. Patient has received any other anti-cancer therapies targeting at CLDN6.
  4. Patient has persisting toxicity of > Grade 1 (NCI CTCAE v5.0) relating to prior anti-cancer therapy with the exceptions of alopecia and endocrine dysfunction which could be managed by replacement therapy.
  5. Patient has active or uncontrolled infections, which require systemic treatment of antibiotics, antivirals, or antifungals, within 2 weeks prior to start of study drug.
  6. Patient has meningeal metastases (symptomatic or asymptomatic), or has symptomatic or uncontrolled brain metastases or spinal cord compression. Patients with asymptomatic brain metastases (longest diameter of brain lesion ≤ 3 cm) can be enrolled only if treated, non-progressive brain metastases and off high-dose steroids (> 20 mg prednisone or equivalent) for at least 4 weeks. If the patient has previously received antiepileptic treatment for central nervous system (CNS) metastases, antiepileptic medications should be discontinued for at least 2 weeks (14 days) prior to start of study drug.
  7. Patient has uncontrolled pleural, peritoneal or pericardial effusion. Asymptomatic and stable effusion could be enrolled if any one of the following criteria is met:

     * If previous imaging indicated the presence of effusion, subsequent imaging shows a reduction, no change, or a slight increase of the effusion volume, and the patient has no effusion related symptom.
     * If puncture drainage or other therapy was performed, reexamination after an interval of 2 weeks at least shows no significant increase of the effusion volume, and the patient has no effusion related symptom.
  8. Patients who have other malignancies requiring treatment within 5 years prior to the first dose of study drug will be excluded, except for radically treated locally curable basal or squamous cell skin cancer, cervical carcinoma in situ, papillary thyroid carcinoma, breast ductal carcinoma in situ and other malignancies with favorable prognosis that have been treated with no relapse within 5 years.
  9. Patients with history of active or chronic corneal and conjunctival diseases; or history of active ocular surface diseases or scarring conjunctivitis; or presence of other clinically significant ocular diseases affecting corneal, conjunctival, or other areas that may impact drug-related ophthalmic toxicity monitoring.
  10. Has a pre-existing clinically significant lung diseases (e.g., interstitial lung disease, non-infectious pneumonitis, pulmonary fibrosis, and severe radiation pneumonitis), with abnormal signs or symptoms, or require treatment.
  11. Patient has severe or unstable cardiac conditions, including:

      * History of congestive heart failure (New York Heart Association Class > 2);
      * History of unstable angina or myocardial infarction within 6 months prior to the first dose of study drug;
      * History of atrial fibrillation, supraventricular arrhythmia, or ventricular arrhythmia within 6 months prior to the first dose of study drug and still in unstable condition and requiring treatment or intervention;
      * QTcF prolongation >470 ms, or risk factors for Torsades de Pointes (such as congenital long QT syndrome, family history of long QT syndrome, unexplained sudden death under the age of 40 years old in first-degree relatives, severe hypokalemia or hypomagnesemia, concomitant use of medication which has known risk of QT prolongation).
  12. Patient with history of cerebrovascular diseases (including but not limited to stroke or transient ischemic attack) within 6 months prior to the first dose.
  13. Patient with uncontrolled hypertension (systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg despite treatment), or uncontrolled diabetes despite treatment.
  14. Patient with active hepatitis B virus (HBV) infection, defined as positive hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb), and HBV deoxyribonucleic acid (DNA) levels higher than 200 IU/mL or 1000 copies/mL.
  15. Patient with active hepatitis C virus (HCV) infection, defined as positive hepatitis C antibody (HCV-Ab) and HCV-ribonucleic acid (RNA) quantified above the upper limit of the normal detection units.
  16. Patient with known history of human immunodeficiency virus (HIV) infection and/or acquired immunodeficiency syndrome.
  17. Patient has major surgery within 2 weeks of first dose of study drug.
  18. Participation in another clinical study with an investigational product administered within 28 days or 5 half-lives (whichever is shorter) prior to receiving the first dose of study drug.
  19. Patient with a known history of hypersensitivity to any components of the study drug, including eribulin and excipients.
  20. Pregnant or breastfeeding women.
  21. Patient with history or evidence of any other clinically significant condition or disease that, in the opinion of the investigator, would be a risk to patient's safety or interfere with the study evaluation, procedures or completion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-12 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Recommended Extension Dose and Recommended Phase 2 Dose (RP2D) | up to 2 years
  Based on the maximum tolerated dose, cumulative safety, and pharmacokinetic data
Incidence and severity of adverse events and serious adverse events | up to 2 years
  Number and percentage of patients with adverse events (AEs), serious adverse events (SAEs), treatment-related adverse events (TRAEs), and dose-limiting toxicities (DLTs) ,according to NCI-CTCAE Version 5.0

SECONDARY OUTCOMES:
Maximum Serum Concentration of PLB-002 (Cmax) | 21 days
  PK assessment
Time of Maximum Serum Concentration of PLB-002(Tmax) | 21 days
  PK assessment
Area under the Serum Concentration-Time curve from the time of dosing to the last measurable concentration (AUClast) for PLB-002 | 21 days
  PK assessment
Area under the Serum Concentration-Time curve from the time of dosing extrapolated to time infinity (AUCinf) for PLB-002 | 84 days
  PK Assessment
Terminal Half-life (t1/2) of Serum PLB-002 | 84 days
  PK Assessment
Apparent volume of distribution during the terminal phase (Vz) of PLB-002 | 84 days
  PK assessment
Clearance (CL) of PLB--002 | 84 days
  PK Assessment
Number of anti-drug antibody (ADA) Positive Participants | up to 2 years
  Immunogenicity will be measured by the number of participants that are ADA positive.
QTc assessment (only applicable for Part 1) | up to 2 years
  To evaluate the effect of different concentrations of PLB-002 on the QTc interval
Objective Response Rate (ORR) | up to 2 years
  Percentage of participants with best response of complete response (CR) or partial response (PR) according to RECIST 1.1
Duration of Response (DOR) | up to 2 years
  Time from CR or PR to objective disease progression or death to any cause
Disease control rate (DCR) | up to 2 years
  Disease control rate (DCR) refers to the percentage of patients achieving CR, PR or SD among all evaluable cases per RECIST v1.1.
Progression Free Survival (PFS) | up to 2 years
  PFS is defined as the time from the start of the treatment until objective disease progression or death from any cause
Overall Survival | up to 2 years
  To assess Overall survival (OS) (only applicable for Part 2)

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Fudan University Shanghai Cancer Center- Gynecology Onc, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center- Phase 1, Shanghai, Shanghai Municipality